CLINICAL TRIAL: NCT06681337
Title: A Clinical Study of the Safety and Efficacy of Universal CAR-T Cells Targeting BCMA and CD19 for the Treatment of Refractory Lupus Nephritis
Brief Title: Universal CAR-T Cell Therapy for Refractory Lupus Nephritis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bioray Laboratories (Industry)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-BRL-302-03
Record Dates: First submitted 2024-11-04; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-09

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA CART + CD19 CART (Experimental): BCMA CART + CD19 CART
  Interventions: Biological: BCMA CART + CD19 CART

INTERVENTIONS:
Biological: BCMA CART + CD19 CART — BCMA CART + CD19 CART

SUMMARY:
This investigator-initiated trial aims to assess the efficacy and safety of combination therapy using universal CAR-T cells targeting BCMA and CD19 in refractory lupus nephritis.

DETAILED DESCRIPTION:
This study is a non-randomized, open-label, single-arm clinical trial designed to assess the efficacy and safety of combination therapy for refractory lupus nephritis using universal CAR-T cells targeting BCMA and CD19.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years; both genders eligible.
* Subjects diagnosed with lupus nephritis.
* Previous treatment outcomes were unsatisfactory.
* Diagnosis of active nephritis type III or IV with or without type V according to 2018 International Society of Nephrology and Society of Renal Pathology (ISN/RPS) criteria.
* NIH Activity Index > 2 and elevated chronicity index.
* Urine protein: creatinine ratio (UPCR) ≥ 1.0 g/g, or 24-hour urine protein ≥ 1.0 g, with or without active urine sediment with red blood cell casts.
* Receiving hormones with or without antimalarials.
* SLEDAI-2K score ≥ 6.
* Antinuclear antibody positive, and/or anti-ds-DNA antibody positive, and/or anti-Smith antibody positive.
* Positive expression of CD19 on B cells in peripheral blood.
* Agrees to use double barrier methods, condoms, oral or injectable contraceptives, or intrauterine devices during the study period and for one year after taking the study medication.
* Provides written informed consent.

Exclusion Criteria:

* History of solid organ transplantation.
* Malignant tumor within the last two years.
* Positive for Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb), with peripheral blood Hepatitis B virus (HBV) DNA detected as positive; positive for Hepatitis C virus antibodies, with peripheral blood Hepatitis C virus RNA detected as positive; positive for Human Immunodeficiency Virus (HIV) antibodies; positive for Cytomegalovirus (CMV) DNA; positive for syphilis.
* Primary immunodeficiency (congenital or acquired).
* Severe cardiac disease.
* History of psychiatric disorders or history of psychotropic drug abuse, with no history of withdrawal.
* Allergic constitution or a history of severe allergies.
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-25 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
AEs | Within 6 months after BCMA CART and CD19 CART infusion
  The total number, incidence, and severity of AE

SECONDARY OUTCOMES:
ORR (CR and PR) | At 6 months after BCMA CART and CD19 CART infusion
  Complete response (CR) was defined as serum creatinine ≤ 1.2 mg/dl or ≤ 125% of baseline value, and urine protein/creatinine ratio < 0.5 or 24-hour urine protein quantification < 0.5 g, and prednisone dose reduction to ≤ 10 mg/d (or equivalent dose). Partial response (PR) was defined as if both serum creatinine and urine protein/creatinine ratio (or 24-hour urine protein quantification) were abnormal before treatment, both items improved by > 30% after treatment, without other indicators of deterioration; if only urine protein/creatinine ratio (or 24-hour urine protein quantification) was abnormal before treatment, the improvement was > 50% after treatment.

OTHER OUTCOMES:
PK/PD | Within 3 months after BCMA CART and CD19 CART infusion
  Changes and duration of CAR gene copy number and CAR-T cell number in peripheral blood after BCMA CART and CD19 CART infusion